CLINICAL TRIAL: NCT05883865
Title: Safety and Efficacy of Fenofibrate in the Treatment of Pregnant Women With Severe Hypertriglyceridemia
Brief Title: Safety Study of Fenofibrate During Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Other Study IDs: IIT-20221208-0197-01
Record Dates: First submitted 2023-05-17; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-04

CONDITIONS: Severe Hypertriglyceridemia During Pregnancy
Keywords: severe hypertriglyceridemia; fenofibrate; pregnancy
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Fenofibrate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — maternal and cord blood, amniotic fluid and breast milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- fenofibrate group: Women with TG level ≥10mM receive fenofibrate micronized capsule（200mg ，qd）or table（160mg ，qd）for at least 1 week during pregnancy.
  Interventions: Drug: Fenofibrate
- negative group: Pregnant women with TG level ≥10mM without fenofibrate treatment.

INTERVENTIONS:
Drug: Fenofibrate — Fenofibrate is orally administrated daily with food for at least 1 week during pregnancy
  Groups: fenofibrate group

SUMMARY:
The purpose of this study is to evaluate the safety of fenofibrate in severe hypertriglyceridemia pregnant women.

DETAILED DESCRIPTION:
Due to changes in various hormone levels during pregnancy, triglyceride (TG) levels will increase physiologically. When TG>10mM, the risk of pancreatitis increases, thereby threaten the maternal and fetal health. Therefore, when TG>10mM, in addition to life interventions such as diet and exercise, drug treatment is required. Fenofibrate is the first-line TG-lowering drug, however, information on its safety during pregnancy is insufficient. According to the instruction, fenofibrate can only be used when the benefits outweigh the risks, that is, dietary control cannot effectively reduce TG (>10g/L) and increase the risk of acute pancreatitis in the mother. This study involves two aspects. On the one hand, it evaluates the effect of fenofibrate on pregnancy outcomes through a retrospective study, and on the other hand, it evaluates its effect on children's growth and development, placental penetration, and milk excretion through a prospective study. 200 pregnant women with TG level>10mM exposed to fenofibrate for more than one week will be recruited. The pregnancy outcomes will be compared to the unexposed women with TG level>10mM. 50 TG level>10mM pregnant women will be enrolled on receive fenofibrate treatment between weeks 24-39 of gestation and delivery for more than one week. According to the mother's wishes, maternal blood, cord blood, amniotic fluid at delivery and breast milk through 7 days after delivery will be collected and for fenofibric acid concentration determination. Moreover, in a one-year follow-up, the physical growth parameters of infants will be collected. The primary endpoint is the effect of fenofibrate on pregnancy outcomes and infant physical growth. The secondary endpoint is placental transfer and milk penetration of fenofibric acid.

ELIGIBILITY:
Inclusion Criteria:

* 20-45 years pregnant women; TG level ≥10mM； Voluntary signed informed consent (prospective study) or voluntary consent to use of medical information (retrospective analysis)

Exclusion Criteria:

* Evidence of decompensated liver disease; Pregnant women with major organ lesions; Has a history of kidney injury, creatinine clearance <50ml/min, positive urine protein (>300mg/L); Combined with other chronic diseases (epilepsy, severe intrahepatic cholestasis of pregnancy, severe preeclampsia, systemic lupus erythematosus, antiphospholipid antibody syndrome); B-ultrasound and other examinations during pregnancy have found fetal malformations, or suggested intrauterine growth retardation, or had birth defects or congenital malformations in the previous pregnancy; Pregnant women are participating in other studies or taking other fibrate lipid-lowering drugs

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women whose TG level is ≥10mM and cannot be decreased by life interventions.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
rate of preterm birth of infants | delivery
Apger score of infants | delivery
body weight of infants | within 1 year after delivery
length of infants | within 1 year after delivery
head circumference of infants | within 1 year after delivery

SECONDARY OUTCOMES:
placental transfer | delivery
  Ratio of fenofibrate concentrations in cord and maternal blood
milk penetration | up to 7 days after delivery
  fenofibrate concentrations in breast milk up to 7 days after delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People's Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No